CLINICAL TRIAL: NCT03462654
Title: Comparison of a Group-delivered and Individually Delivered Lifestyle-integrated Functional Exercise (LiFE) Program in Older Persons
Brief Title: Comparison of a Group-delivered vs. Individually Delivered 'LiFE' Program
Acronym: LiFE-is-LiFE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Heidelberg University (Other)
Collaborators: Robert Bosch Gesellschaft für Medizinische Forschung mbH (RBMF) (Other); University of Ulm (Other); Universitätsklinikum Hamburg-Eppendorf (Other); German Federal Ministry of Education and Research (Other Government)
Responsible Party: Principal Investigator, Carl-Philipp Jansen, Post-Doctoral Research Assistant, Heidelberg University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 01GL1705A-D
Record Dates: First submitted 2018-02-26; First posted 2018-03-12 (Actual); Last update posted 2022-08-25 (Actual); Status verified 2022-08

CONDITIONS: Fall Prevention; Exercise
Keywords: Health promotion; Behaviour change; Physical activity; Fall prevention
MeSH Terms: conditions — Motor Activity

STUDY DESIGN:
Intervention Model Description: Participants will be randomized into either the iLiFE or gLiFE arm of the study.
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- individual LiFE (iLiFE) (Active Comparator): In iLiFE, LiFE activities to increase strength, improve balance, and promote physical activity as well as habitualization strategies are introduced and taught in 7 highly individualized, one-to-one home visits.
  Interventions: Behavioral: iLiFE
- group LiFE (gLiFE) (Experimental): In gLiFE, the same LiFE activities as performed in iLiFE are introduced and taught in 7 group sessions with 8 to 12 participants. Implementation and habitualization strategies will be addressed within the group setting, making use of group dynamics and processes.
  Interventions: Behavioral: gLiFE

INTERVENTIONS:
Behavioral: iLiFE — In the individual LiFE (iLiFE), the program is taught in seven visits in the individuals' homes within eleven weeks. Participants are supervised in a face to face situation by one qualified trainer (physiotherapist or sports scientist). Each home visit takes between 1 and 1.5 hours. A total of five balance exercises, seven strength exercises for the lower extremities, and two exercises to increase physical activity are taught. In addition to the home visits, all participants receive two 'booster telephone calls' within the remaining weeks until the 6-month follow-up assessments.
  Arms: individual LiFE (iLiFE)
Behavioral: gLiFE — The group-based LiFE (gLiFE) program consists of seven group sessions (n = 8-12 participants) which are held over the course of eleven weeks, with a maximum duration of 2 hours per session. Each session is led by two qualified trainers (physio therapists or sports scientists), i.e., one main and one co-trainer. In all group sessions, trainers will teach the participants how to perform and integrate the LiFE program, i.e., LiFE balance and strength activities into their daily routines. After the group sessions have ended, participants will receive two 'booster telephone calls' within the remaining weeks until the 6-month follow-up assessments.
  Arms: group LiFE (gLiFE)

SUMMARY:
In the Lifestyle-Integrated Functional Exercise (LiFE) program, exercises to increase strength and improve balance are embedded into daily life activities. Recurring daily activities and tasks are used as prompts for these exercises so that they are performed multiple times per day. However, implementing the original LiFE program includes high financial requirements and human resources as it comprises one-to-one supervision of participants. Therefore, it is investigated whether implementing LiFE in groups (gLiFE) is not inferior to the individually delivered LiFE (iLiFE) in terms of reducing falls per physical activity. In addition, gLiFE is expected to be more cost-effective as compared to iLiFE. In a multicenter non-inferiority trial, 300 participants aged 70 years or older with confirmed fall risk will be randomized into either the iLiFE or gLiFE arm of the study. Both arms will undergo the same strength and balance exercises and habitualization strategies as described in the LiFE program, however, based on different approaches of delivery (i.e., group vs. individual).

DETAILED DESCRIPTION:
The "Lifestyle-integrated Functional Exercise" (LiFE) program aims to promote safe indoor and outdoor mobility. It differs from classical exercise programs in that it trains and encourages participants to embed up to 15 balance and strength exercises into daily recurring tasks performed as part of the daily life routine. The LiFE program simultaneously aims at preventing falls and promoting an active lifestyle in older adults. As LiFE requires 1:1 supervision by trainers who administer LiFE exercises during seven visits in the participants' homes, it is both time consuming and resource intensive and therefore not suitable for widespread implementation. Hence, the aim of this study is to compare a group-delivered LiFE intervention (gLiFE) with the original LiFE intervention (iLiFE). More specifically, gLiFE is tested for its non-inferiority compared to iLiFE in terms of:

* Effectiveness: The gLiFE program is not less efficacious than the established iLiFE program in terms of reducing fall incidence expressed as number of falls per amount of physical activity (e.g., steps).
* Retention rate: The gLiFE program does not result in a lower intervention retention rate (i.e., percentage of the sample completing the 6-month and 12-month follow-up assessment) as compared to the iLiFE program.
* Implementation: Delivering the gLiFE program is less costly and more cost-effective than delivering the iLiFE program.

In a multicenter non-inferiority trial, participants (n = 300; > 70 years; confirmed fall or high risk of falling) will be randomized into either the individual iLiFE (seven home visits) or gLiFE (groups up to twelve persons; seven group sessions).

ELIGIBILITY:
Inclusion Criteria:

* Aged 70 years or older
* Speaks German language
* Able to read newspaper
* Able to walk 200 meters with or without walking aid
* Home-dwelling
* Two or more falls in the past 12 months OR one injurious fall in the past 12 months OR subjective decline in balance and strength in the past 12 months together with Timed Up-and-Go time >13.5 seconds
* Available for intervention participation for 11 weeks

Exclusion Criteria:

* Cognitive impairment (MoCA <23)
* Current participation in an organised exercise class >1 per week in the past 3 months
* Moderate to vigorous-intensity physical activity ≥150 min/week in the past 3 months
* Medical conditions:

  1. Heart failure New York Heart Function Assessment (NYHA) class III and IV
  2. Recent cerebrovascular accident (<6 months)
  3. Parkinson's disease
  4. On active cancer treatment (last 6 months)
  5. Chronic Obstructive Pulmonary Disease (COPD) Gold class III and IV
  6. Unstable lower limb fracture
  7. Amputated lower extremity (-ies)
  8. Acute treatment of depression
  9. Uncontrolled resting blood pressures of a systolic >160 or diastolic >100 or higher

Min Age: 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 310 (Actual)
Dates: Start 2018-04-05 (Actual); Primary Completion 2020-08-05 (Actual); Study Completion 2020-09-30 (Actual)

PRIMARY OUTCOMES:
Fall incidence expressed as number of falls per amount of physical activity | Change; baseline, 6 months, 12 months
  Falls are assessed using a fall calendar; Physical activity is assessed using activPAL accelerometers
Cost-effectiveness of iLiFE and gLiFE | Change; baseline, 6 months, 12 months
  Incremental Cost-Effectiveness Ratios (ICERs) of delivering iLiFE and gLiFE

SECONDARY OUTCOMES:
Accelerometer-collected physical activity (duration) | Change; baseline, 6 months, 12 months
  Duration of sedentary, active, and walking time during 7 days as assessed using 'activPAL' activity monitors
Accelerometer-collected physical activity (percentage) | Change; baseline, 6 months, 12 months
  Percentage of sedentary, active, and walking time during 7 days as assessed using 'activPAL' activity monitors
Accelerometer-collected physical activity (intensity) | Change; baseline, 6 months, 12 months
  Intensity of sedentary, active, and walking time during 7 days as assessed using 'activPAL' activity monitors
Adherence to LiFE activities | Monthly; starting from first iLiFE or gLiFE participation until the date of the 12 month follow-up
  Exercise Adherence Rating Scale (EARS) filled out every month in a calendar
Self-reported function and disability | Change; baseline, 6 months, 12 months
  Late-Life Function and Disability Instrument (LLFDI)
Static balance (a) | Change; baseline, 6 months, 12 months
  8 Level Balance Scale
Static balance (b) | Change; baseline, 6 months, 12 months
  Instrumented Tandem Stance
Gait speed | Change; baseline, 6 months, 12 months
  instrumented walking test (4m and 7m walk at usual and fast pace)
Functional leg strength (a) | Change; baseline, 6 months, 12 months
  Instrumented 30 second Chair Stand
Functional leg strength (b) | Change; baseline, 6 months, 12 months
  Instrumented Timed Up-and-Go
Handgrip strength | Change; baseline, 6 months, 12 months
  JAMAR dynamometer
Cognitive status | Change; baseline, 6 months, 12 months
  Montreal Cognitive Assessment Tool (MoCA)
Balance confidence | Change; baseline, 6 months, 12 months
  Activities-specific Balance Confidence Scale (ABC-Scale)
Fear of falling | Change; baseline, 6 months, 12 months
  Short Falls Efficacy Scale-International (Short FES-I)
Health status (a) | Change; baseline, 6 months, 12 months
  EQ-5D-5L
Health status (b) | Change; baseline, 6 months, 12 months
  EQ-VAS
Health-related resource use | Change; baseline, 6 months, 12 months
  questionnaire for the use of medical and non-medical services in old age (FIMA)
Depressive Symptoms | Change; baseline, 6 months, 12 months
  10 Item Center for Epidemiological Studies - Depression (CES-D-10)
Subjective age | Change; baseline, 6 months, 12 months
  Subjectively felt age in years
Habit strength | Change; baseline, 6 months, 12 months
  Self-Report Behavioural Automaticity Index (SRBAI)
Motivational quality | Change; baseline, 12 months
  Behavioural Regulation in Exercise Questionnaire (BRE-Q-3)
Health Action Process Approach (HAPA) - Int | Change; baseline, 6 months, 12 months
  Intention (2 items, 6-point Likert scale)
Health Action Process Approach (HAPA) - SE | Change; baseline, 6 months, 12 months
  Self-efficacy (6 items, 6-point Likert scale)
Health Action Process Approach (HAPA) - ACP | Change; baseline, 6 months, 12 months
  Action and coping planning (6 items, 6-point Likert scale)
Health Action Process Approach (HAPA) - IAC | Change; baseline, 6 months, 12 months
  Individual action control (3 items, 6-point Likert scale)
Social support | Change; baseline, 6 months, 12 months
  Loneliness Scale
Group cohesion | Change; baseline, 6 months, 12 months
  Kohäsion im Team von Freizeit- und Gesundheitssportgruppen Scale (German)
Evaluation of the LiFE program | Change; after the last intervention session, 6 months, 12 months
  10 questions regarding quality and acceptance of as well as satisfaction with the program (6-point Likert scale)

CONTACTS AND LOCATIONS:
Overall Officials: Michael Schwenk, PhD, Principal Investigator — Network Aging Research
Locations (2):
- Germany (2):
  - Heidelberg University, Network Aging Research, Heidelberg
  - Robert Bosch Hospital, Klinik für Geriatrische Rehabilitation, Stuttgart

REFERENCES:
- [Derived] Dams J, Gottschalk S, Schwenk M, Nerz C, Becker C, Klenk J, Jansen CP, Konig HH. Budget impact analysis of a Lifestyle-integrated Functional Exercise (LiFE) program for older people in Germany: a Markov model based on data from the LiFE-is-LiFE trial. BMC Geriatr. 2024 Feb 23;24(1):186. doi: 10.1186/s12877-024-04802-y. PMID 38395743
- [Derived] Nerz C, Kramer-Gmeiner F, Jansen CP, Labudek S, Klenk J, Becker C, Schwenk M. Group-Based and Individually Delivered LiFE: Content Evaluation and Predictors of Training Response - A Dose-Response Analysis. Clin Interv Aging. 2022 Apr 27;17:637-652. doi: 10.2147/CIA.S359150. eCollection 2022. PMID 35509348
- [Derived] Jansen CP, Nerz C, Labudek S, Gottschalk S, Kramer-Gmeiner F, Klenk J, Dams J, Konig HH, Clemson L, Becker C, Schwenk M. Lifestyle-integrated functional exercise to prevent falls and promote physical activity: Results from the LiFE-is-LiFE randomized non-inferiority trial. Int J Behav Nutr Phys Act. 2021 Sep 3;18(1):115. doi: 10.1186/s12966-021-01190-z. PMID 34479573
- [Derived] Reicherzer L, Kramer-Gmeiner F, Labudek S, Jansen CP, Nerz C, Nystrand MJ, Becker C, Clemson L, Schwenk M. Group or individual lifestyle-integrated functional exercise (LiFE)? A qualitative analysis of acceptability. BMC Geriatr. 2021 Feb 1;21(1):93. doi: 10.1186/s12877-020-01991-0. PMID 33522904
- [Derived] Jansen CP, Nerz C, Kramer F, Labudek S, Klenk J, Dams J, Konig HH, Clemson L, Becker C, Schwenk M. Comparison of a group-delivered and individually delivered lifestyle-integrated functional exercise (LiFE) program in older persons: a randomized noninferiority trial. BMC Geriatr. 2018 Nov 6;18(1):267. doi: 10.1186/s12877-018-0953-6. PMID 30400832
- See also: Project homepage — http://www.life-alltagsuebungen.de